CLINICAL TRIAL: NCT01616160
Title: An Open-label Study to Identify Molecular Markers of Steroid Resistance in Nasal Polyposis Before and Following Treatment With Mometasone Furoate (MFNS) 2 Sprays/Nostril (100 mcg/Nostril) Twice Daily for 4 Weeks.
Brief Title: An Open-label Study to Identify Molecular Markers of Steroid Resistance
Acronym: MERK2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit additional subjects.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Daniel Hamilos MD, Principle Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012P000387
Record Dates: First submitted 2012-05-30; First posted 2012-06-11 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Nasal Polyps
Keywords: Nasal polyps
MeSH Terms: conditions — Nasal Polyps | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nasal polyps subjects (Experimental): 24 subjects with nasal polyps. Intervention: Each subject will receive Nasonex (mometasone furoate) 2 spray per nostril twice daily for 4 weeks.
  Interventions: Drug: mometasone furoate

INTERVENTIONS:
Drug: mometasone furoate — 2 sprays/nostril BID
  Other Names: Nasonex

SUMMARY:
Aim 1: To assess steroid sensitivity to mometasone furoate (MF) in cultured nasal polyp explant tissue in vitro.

Aim 2: To assess steroid sensitivity in vivo in each subject by comparing symptom scores, nasal endoscopic findings before and following 4 weeks of treatment with mometasone furoate nasal spray (MFNS) and by comparing tissue immunohistology in NP biopsies pre- and post-treatment withA MFNS.

Aim 3: To characterize the molecular signature of gene mRNA expression in "steroid-sensitive" and "steroid-resistant" NP using microarray on NP tissue pre- and post-MFNS treatment.

Hypothesis 1: Genes that regulate apoptosis are dysregulated in nasal polyp (NP) inflammatory cells, epithelial cells and smooth muscle actin myofibroblasts leading to persistence of inflammatory cell infiltration and abnormal epithelial and myofibroblast cellular proliferation. These can be corrected by mometasone. Apoptosis-regulating genes that cannot be corrected by mometasone are upregulated in steroid-resistant NP.

Elucidation of this dysregulation may prove insightful in understanding the mechanism of action of mometasone in NP and identifying potential molecular targets that will increase steroid sensitivity or, conversely, overcome steroid resistance.

Hypothesis 2: There is a molecular signature of gene expression in NP that signifies steroid sensitive NP (SS-NP). This signature is altered in steroid resistant NP (SR-NP).

Elucidation of differences in the molecular signature of SS-NP versus SR-NP before and after treatment with mometasone furoate (MFNS) will provide novel insight into treatment of NP with steroids.

DETAILED DESCRIPTION:
Visit 1: Baseline evaluation and nasal endoscopy

At this visit, each subject will sign an informed consent, the subject's eligibility for the study will be confirmed, a medical history will be obtained, the subject will undergo a physical examination and nasal endoscopy. A urine pregnancy test will be performed on all females of childbearing potential. NP size will be recorded using the NP scoring system (see below).

Allergy skin testing will only be performed if it has not been done in the past 3 years.

Visit 2: Pre-treatment nasal polyp (NP) biopsies

At this visit, each subject will undergo the pre-treatment NP biopsies. The biopsies will be obtained by Dr. Eric Holbrook at Massachusetts Eye & Ear Infirmary, located adjacent to MGH.

Visit 3: Initiation of treatment with MFNS

At this visit, each subject will have a nasal speculum examination to confirm that there is no residual bleeding from the NP biopsies. Then, the subject will be given a 4 week supply of MFNS (Nasonex ®) and be instructed to take 2 sprays/nostril BID. Subjects will be given a NP symptom diary and instructed to record NP symptoms daily for 4 weeks.

Each subject will be assigned a unique number (screening or baseline number) for identification purposes. Under no circumstances will a patient be assigned more than one allocation number. The Nasonex bottles will be dispensed from the MGH Research Pharmacy.

Visit 4: On-treatment NP biopsy

At this visit, each subject will undergo the on-treatment NP biopsies. The biopsies will be obtained by Dr. Eric Holbrook at Massachusetts Eye & Ear Infirmary, located adjacent to MGH. The subject will be asked to withhold Nasonex treatment for 48 hours following this biopsy.

Visit 5: Post-biopsy Exam At this visit, each subject will have a nasal speculum examination to confirm that there is no residual bleeding from the NP biopsies. If bleeding has ceased, the subject will resume Nasonex treatment.

Visit 5 6: Final visit and nasal endoscopy

At this visit, each subject will return their used and unused bottles of Nasonex and submit their NP symptom diary and undergo a nasal endoscopy. NP size will be recorded using the NP scoring system (see below). Subjects will also complete a global assessment of efficacy of MFNS for their NP symptoms.

EXPERIMENTAL PROCEDURES:

Pre-biopsies explant cultures: we will obtain NP biopsies for in vitro explant culture before steroid treatment from each patient. We will culture the explants in MF at 0, 10-9, 10-8, 10-7, 10-6, 10-5M and analyze inflammatory cell infiltrate and steroid sensitivity based on induction of apoptosis (activated caspase-3 expression) in inflammatory cell subsets, alpha-smooth muscle cell actin+ myofibroblasts and epithelial cells. Each condition will be performed in duplicate so that one sample can be processed for IHC and one for microarray.

Explant cultures: NP explants will be cultured in minimal essential medium for 24 hours at 37oC using flat-bottom tissue culture plates. Following 24 hours in culture, 1 explant per condition will be processed for IHC and 1 for microarray. We will also save culture supernatant from each explant condition for confirmation of important differences in protein production, based on data from the IHC and microarrays.

Immunohistochemistry (IHC) and confocal laser immunofluorescence microscopy (CLM): Frozen NP samples from SS-NP and SR-NP patients before and after MFNS treatment will be analyzed by immunofluorescence confocal laser microscopy (IF-CLM) for T lymphocyte (CD3 and CD4), MBP+ eosinophils, alpha-smooth muscle actin (marker of activated myofibroblasts, monoclonal, R & D Systems, Inc.) and cleaved caspase-3 (polyclonal, CST, Beverly, MA). The number of inflammatory cells of each type and cleaved caspase-3 positive and negative cells of each type will be counted by two observers blinded to treatment and order of collection. A similar quantification of epithelial staining for PCNA (a marker of epithelial cell proliferation) and cleaved caspase-3 will be performed using semiquantitative grading of extent and intensity of staining as in our previous studies. The intensity and distribution of immunostaining will be quantified on a semi-quantitative grading scale of: 0 = absent staining, 1 = mild diffuse or moderate patchy staining; 2 = moderate diffuse staining; 3 = intense diffuse staining in the epithelium, stroma and glands by 2 independent observers.

Histologic steroid-sensitive and steroid-resistant phenotype designation: Designation of NP subjects as histologically "steroid-sensitive" or "steroid-resistant" will be based on the following measures pre- and 1-week post-treatment with MFNS:

1. extent of reduction in NP eosinophils improvement in NP inflammation,
2. extent of induction of apoptosis in eosinophils, T lymphocytes and epithelial cells,
3. extent of suppression of inflammatory gene expression based on microarray analysis.

Subjects will be ranked in order from most sensitive to least sensitive to treatment. Linear regression will be used to examine correlations between these independent continuous variables.

Microarray analysis: microarray analysis will be used to assess global gene mRNA expression and also capture information on pro- and anti-apoptotic gene expression in "steroid sensitive" (SS-NP) and "steroid resistant" SR-NP biopsies obtained before and 1 week following treatment with intranasal mometasone furoate (MFNS). RNA isolation for microarray is done using the Arcturus picopure RNA isolation system. Plastic LCM collecting caps are incubated at 42oC for 30 minutes in 25 microliter of the kit's GITC-containing extraction buffer, centrifuged briefly to collect the extracted solution, then frozen at -80oC. Samples are thawed and pooled prior to purification on picopure RNA columns, and genomic DNA is removed via RNAse-free DNAse (Qiagen, Hilden, GmbH) digestion on the columns. Total cellular RNAs from each column are eluted in 11 microliter of elution buffer and used for preparation of the RNA-Seq library, or converted into cDNA-for the QRTPCR assay, using a 20 microliter total reaction volume via the standard superscript III (Invitrogen, Carlsbad, CA) protocol. We also have microarray data from 8 healthy control middle turbinates obtained in a previous study that will be used for comparison of gene expression to nasal polyps.

RNA will be purified from one NP biopsy per patient using the ArrayPure™ Nano-scale RNA Purification Kit, (EPICENTRE Biotechnologies, Madison, WI) which includes ScriptGuard™ RNase Inhibitor to maintain the integrity of purified RNA. Purified RNA quality will be checked using RNA Nano Analysis (Agilent Bioanalyzer, Quantum Analytics, Inc., Foster City, CA). The lower limit sensitivity is 200 pg/ml, allowing us to verify the quality of RNA extracted from about 1250 cells.

QRTPCR: Genes that are differentially expressed by RNA expression profiling will be further investigated by quantitative real-time RT-PCR from a separate small sample of purified RNA from each tissue compartment. RT-PCR will be performed using the Multiplex MX3000P quantitative RT-PCR system (Stratagene, La Jolla, CA). Baseline gene expression will be quantified by QRTPCR relative to GAPDH using the delta-delta Ct (2-∆∆) method. Forward and reverse primers will be selected based on primerbank software (http://pga.mgh.harvard.edu/primerbank/). To confirm gene-expression within tissues we will use immunohistochemistry as in previous studies.

ELIGIBILITY:
Inclusion Criteria:

- The subject must fulfill all of the following conditions or characteristics to be considered for enrollment:

1. Male or female between ages 21 - 70 years residing in the Boston area
2. History of chronic rhinosinusitis (symptoms for at least 3 months). Subject must have two or more of the following:

   * Facial pain/pressure or headache
   * Nasal congestion
   * Anterior or posterior nasal drainage
   * Hyposmia/anosmia
3. Abnormal CT scan in at least 2 sinuses areas within 3 months
4. Evidence of bilateral polyps or polypoid mucosa (on nasal endoscopy) with minimum polyp/polypoid score of 4 (see scoring system below).

   Exclusion Criteria:
   * 4. History of suggestive of immunodeficiency (i.e. those who have had > one pneumonia in the past 12 months or those with known immune deficiency).
5. History of cystic fibrosis, Kartagener's syndrome, immotile cilia syndrome, hypogammaglobulinemia or bleeding disorder
6. URI within six weeks prior to enrollment
7. Intranasal cocaine use
8. Pregnancy (if applicable
9. History of fainting

   MEDICATION EXCLUSIONS prior to NP biopsies:
10. Use of prescription blood thinners
11. Use of systemic glucocorticoids for two weeks prior to enrollment
12. Use of intranasal corticosteroids and anticholinergics for three days prior to enrollment
13. Use of an antibiotic for three days prior to enrollment
14. Use of antihistamines for one week prior to enrollment

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2017-01 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hamilos, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nasal Polyps Subjects: Intervention: Each subject will receive Nasonex (mometasone furoate) 2 spray per nostril twice daily for 4 weeks.
  mometasone furoate: 2 sprays/nostril BID
Period: Overall Study
Arm/Group | Nasal Polyps Subjects
Started | 11
Completed | 9
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nasal Polyps Subjects
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Steroid Sensitivity in Vivo Symptom Scores - Trouble With Sense of Smell
Description: To assess steroid sensitivity in subjects comparing Trouble with sense of smell symptom scores before and following 4 weeks treatment with mometasone furoate nasal spray (MFNS). Trouble with sense of smell measured on 0 to 4 scale ( 0 = no trouble with smell; 4 = severe trouble with smell). The outcome is the difference in mean score (Post - Pre). A negative difference would indicate patients had less trouble with sense of smell at the end of the study.
Time Frame: Change between pre- and post-treatment symptom score after 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Nasal Polyps Subjects: Intervention: Each subject received Nasonex (mometasone furoate) 2 spray per nostril twice daily for 4 weeks.
  mometasone furoate: 2 sprays/nostril twice daily
Arm/Group | Nasal Polyps Subjects
Number analyzed (Participants) | 9
scores on a scale | -0.9 (1.66)

2. Primary Outcome: Change in Steroid Sensitivity in Vivo Nasal Endoscopy Polyp Scores
Description: To assess steroid sensitivity in subjects comparing nasal endoscopy polyp score before and following 4 weeks treatment with mometasone furoate nasal spray (MFNS). Nasal endoscopic polyp score measured on 0 to 4 scale ( 0 = no nasal polyp; 1 = polyp in the middle meatus, not below the inferior border of the middle turbinate (MT); 2 = polyp below the inferior border of the MT but not touching the inferior turbinate (IT); 3 = polyp below the inferior border of the MT and touching the IT; 4 = polyp to or below the lower border of the IT). The outcome is the difference in mean score (Post - Pre). A negative difference would indicate that patients had a reduction in nasal polyp size at the end of the study.
Time Frame: Change between pre- and post-treatment symptom score after 4 weeks of treatment
Population: Each subject received Nasonex (mometasone furoate) 2 spray per nostril twice daily for 4 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nasal Polyps Subjects
Number analyzed (Participants) | 9
units on a scale
  Right nasal polyp | 0 (1.07)
  Left nasal polyp | -0.25 (1.66)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Nasal Polyps Subjects
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes